CLINICAL TRIAL: NCT05500664
Title: The Effect of Aromatherapy on Anxiety in Patients Undergoing Genicular Nerve Radiofrequency for Painful Knee Osteoarthritis
Brief Title: The Effect of Aromatherapy on Anxiety in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00202205
Record Dates: First submitted 2022-01-02; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — lavender oil

STUDY DESIGN:
Intervention Model Description: We hypothesized that the use of lavender aromatherapy before surgery would reduce preintervntion of radiofrequency anxiety as assessed by the Speilberger State-Trait Anxiety Inventory (STAI) questionnaire
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lavender (Active Comparator): three drops of the designated lavender will be placed on a 2-inch by 2-inch impermeable, backed gauze pad and patient was asked to inhale deeply for 5 minutes
  Interventions: Drug: Lavender Oil
- Control (No Intervention)

INTERVENTIONS:
Drug: Lavender Oil — three drops of the designated lavender will be placed on a 2-inch by 2-inch impermeable, backed gauze pad and patient was asked to inhale deeply for 5 minutes
  Arms: Lavender

SUMMARY:
Preoperative anxiety is considered a potential and preventable risk factor for postoperative complications.

DETAILED DESCRIPTION:
Alot of patients face fear from intervention such as radiofrequency. The group of patients with chronic knee osteoarthritis already and mostly have some sore of psychological upset, radiofrequency itself , even in the presence of good periinterventional local anesthetic infiltration, the patients suffer pain and stress. It is well evidenced that aromatherapy specially with Lavender oil offers some sort of anxiety alleviation, pain alleviation and protection against postoperative nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

* adult patients with knee osteoarthritis
* scheduled for genicular nerve radiofrequency

Exclusion Criteria:

* Allergy to lavender
* psychological disorders
* upper respiratory tract illness

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
change of Speilberger State-Trait Anxiety Inventory | preintervention, 15 minutes postintervention
  change of Speilberger State-Trait Anxiety Inventory , There are 20 questions (I feel calm, secure, tense, strained, at ease, upset, am presently worrying over possible misfortunes, satisfied, frightened, uncomfortable, self-confident, nervous, jittery, indecisive, relaxed, content, worried, confused, steady and pleasant) where people rate their anxiety from one (not at all) to four (very much so), and scores range from 20 to 80. low anxiety is 20 to 37, moderate anxiety is 38 to 44, and high anxiety is 45 to 80.

SECONDARY OUTCOMES:
change of Pain visual analog scale | Preintervention, 15 minutes postintervention
  change of Pain visual analog scale, Scale from 0 ( no pain ) up to 10 (worst experienced pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided